CLINICAL TRIAL: NCT00896662
Title: Analysis of Dendritic Phenotype and Function of Patients Receiving VEGF-Trap on VGFT-ST-0202
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey A. Sosman, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC PHI 0433; VU-VICC-PHI-0433; VU-IRB-040852
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoma; Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage IV marginal zone lymphoma; nodal marginal zone B-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Immunologic Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 50cc of peripheral blood will be collected in CPT tubes for mononuclear cell isolation and 10cc in SST tubes for plasma collection.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: immunologic technique — immunologic technique
Other: laboratory biomarker analysis — laboratory biomarker analysis
Other: pharmacological study — pharmacological study

SUMMARY:
RATIONALE: Studying the dendritic cells in samples of blood from patients with cancer receiving aflibercept may help doctors learn about the effect of aflibercept on dendritic cells.

PURPOSE: This laboratory study is evaluating dendritic cells in patients with advanced solid tumors or non-Hodgkin lymphoma receiving aflibercept on clinical trial VGFT-ST-0202.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the effect of in vivo aflibercept on the presence of different populations of dendritic cells (DC) and immature cells (ImC) in the peripheral blood of cancer patients by characterizing the time course (kinetics) of the improvement in antigen presenting cell (APC) phenotype (decline in DC/ImC ratio) occurring early and late after aflibercept administration.
* Evaluate the effect of aflibercept administration on DC function based on ability to stimulate antigen specific proliferative (allogeneic and tetanus toxoid) and cytolytic T cell responses (influenza) by characterizing the time course (kinetics) of the improvement in APC function occurring early and late after aflibercept administration.
* Explore the relationship of baseline aflibercept level and host APC phenotype.

OUTLINE: This is a multicenter study.

Patients undergo phlebotomy and blood collection at baseline and on days 15, 29, and 57. Samples are analyzed for dendritic cell phenotype, subpopulations, maturation status, and function in terms of ability to activate autologous T cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced solid tumor or non-Hodgkin lymphoma and enrolled on clinical trial VGFT-ST-0202
* Hemoglobin ≥ 10 g/dL
* Willing to undergo phlebotomy

Exclusion Criteria:

* none listed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 25 patients; three at each dose level achieved in order to gain additional information regarding safety, pharmacokinetics, and biological effect of VEGF Trap given intravenously.
  Patients with a solid tumor and is consented and eligible for enrollment onto VGFT-ST-0202. Patients who are willing to undergo phlebotomy prior to treatment, and 14 and 28 and 57 days following initial dose of VEGF-Trap. Patients with an Hgb ≥10gm at the time of blood draw.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Effect of in vivo aflibercept on the presence of different populations of dendritic cells (DC) and immature cells (ImC) | at days 15, 29 and 64
Effect of aflibercept administration on DC function based on ability to stimulate antigen specific proliferative (allogeneic and tetanus toxoid) and cytolytic T cell responses (influenza) | at days 15, 29 and 64
Correlation of aflibercept level with host antigen presenting cell phenotype at baseline | at days 15, 29 and 64

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Sosman, MD, Study Chair — Vanderbilt-Ingram Cancer Center